CLINICAL TRIAL: NCT03567746
Title: Efficacy and Safety of Underwater Endoscopic Mucosal Resection Versus Conventional Endoscopic Mucosal Resection for the Treatment of Large Non-pedunculated Colonic Lesions. Multicentric Randomized Controlled Trial
Brief Title: Underwater EMR vs. Conventional EMR for Large Non-pedunculated Colonic Polyp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEMR
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Colonic Polyp
Keywords: Colonic Polyp; Endoscopic mucosal resection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Underwater EMR (Experimental): The patients randomized in this arm will be treated by endoscopic resection assisted by the filling of the colonic lumen using water instead of air and avoiding the formation of a submucosal cushion
  Interventions: Procedure: Underwater EMR
- Conventional EMR (Active Comparator): The patients randomized in this arm will be treated by endoscopic resection following the traditional technique. It means, by assistance of selective submucosal saline injection to create a submucosal cushion below the polyp.
  Interventions: Procedure: Conventional EMR

INTERVENTIONS:
Procedure: Underwater EMR — Polypectomy is performed under full water emersion avoiding the use of submucosal injection.
  Arms: Underwater EMR
Procedure: Conventional EMR — It will be performed in a 2-step procedure. First the formation of a submucosal injection underneath the polyp to create a submucosal safety cushion. Then EMR is performed with a polipectomy snare.
  Arms: Conventional EMR

SUMMARY:
To analyse the efficacy and safety of two standard methods of endoscopic mucosal resection (EMR) for large non-pedunculated colorectal polyps, the investigators will compare submucosal injection-assisted endoscopic mucosal resection (SEMR) versus underwater endoscopic mucosal resection, without submucosal injection (UEMR).

DETAILED DESCRIPTION:
Underwater endoscopic mucosal resection (UEMR) emerges as a variant of traditional resection, in which a submucosal cushion formation is not necessary. This technique was described in 2012 by Kenneth Binmoeller based on the physical floating effect of colonic mucous membrane by filling the colonic lumen using water instead of air. This "floating effect" conditions the natural separation of the colonic wall layers, allowing the distension of the submucosal space without the need to inject substances into it. On the other hand, performing resection in liquid medium conditions could drive the benefit of heat dissipation caused by the current, which would reduces thermal damage caused to the tissues.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged >18 years, diagnosed with a large (>=20 mm) non-pedunculated colonic polyp, who consent to endoscopic mucosal resection of the polyp and willing to participate in this study.

Exclusion Criteria:

* Polyps showing signs of deep submucosal invasion
* Inflamatory bowel disease with signs of activity
* Known or suspected pregnancy
* Patients unable or unwilling to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Lesion recurrence rate | 1 year
  Presence of polyp tissue at the same site as the original lesion (adenoma or sessile serrated polyp)

SECONDARY OUTCOMES:
Technical success rate | 1 hour
  Complete removal of polypoid tissue during the procedure
Incidence of Treatment-Emergent Adverse Events | 1 year
  Incidence of Treatment-Emergent Adverse Events (delated hemorrhage, perforation, hospital admission)
En bloc Resection rate | 1 hour
  Rate of endoscopic mucosal resection in one piece during the procedure
Procedure time | 1 hour
  Time in minutes for the endoscopic mucosal resection
Number of fragments | 1 hour
  Number of fragments of the endoscopic mucosal resection
Lesion size | 1 hour
  Size of the lesion in millimeters
Thermal artecfacts | 1 hour

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital del Mar. Parc de Salut Mar, Barcelona
  - Hospital General Universitario de Ciudad Real, Ciudad Real

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez Sanchez J, Alvarez-Gonzalez MA, Pellise M, Coto-Ugarte D, Uchima H, Aranda-Hernandez J, Santiago Garcia J, Marin-Gabriel JC, Riu Pons F, Nogales O, Carreno Macian R, Herreros-de-Tejada A, Hernandez L, Patron GO, Rodriguez-Tellez M, Redondo-Cerezo E, Sanchez Alonso M, Daca M, Valdivielso-Cortazar E, Alvarez Delgado A, Enguita M, Montori S, Albeniz E. Underwater versus conventional EMR of large nonpedunculated colorectal lesions: a multicenter randomized controlled trial. Gastrointest Endosc. 2023 May;97(5):941-951.e2. doi: 10.1016/j.gie.2022.12.013. Epub 2022 Dec 23. PMID 36572129